CLINICAL TRIAL: NCT03412006
Title: A Randomized, Double-blind, Multicenter Study to Assess the Efficacy and Safety of a 6 Month Oral Treatment With the Chymase Inhibitor BAY 1142524 at a Dose of 25 mg BID in Comparison to Placebo on Top of Standard of Care in Patients With Type II Diabetes and a Clinical Diagnosis of Diabetic Kidney Disease
Brief Title: A Double-blind Study to Investigate Efficacy, Safety and Tolerability of BAY1142524 in Patients With Type II Diabetes and a Clinical Diagnosis of Diabetic Kidney Disease
Acronym: CADA DIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18933; 2017-000656-26 (EudraCT Number)
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Kidney Disease
Keywords: type II diabetes; diabetic kidney disease
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — fulacimstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fulacimstat (BAY1142524) (Experimental): Patients have to have a clinical diagnosis of diabetic kidney disease and have to be treated with standard of care for this condition
  Interventions: Drug: Fulacimstat (BAY1142524)
- Placebo (Placebo Comparator): Patients have to have a clinical diagnosis of diabetic kidney disease and have to be treated with standard of care for this condition
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fulacimstat (BAY1142524) — 25 mg BAY1142524 are given twice daily over a treatment period of 6 months
  Arms: Fulacimstat (BAY1142524)
Drug: Placebo — Matching placebo tablets are given twice daily over a treatment period of 6 months
  Arms: Placebo

SUMMARY:
The purpose of the trial is the analysis of safety and efficacy of the chymase inhibitor BAY1142524 at a dose of 25 mg BID in comparison to placebo using a 6 months treatment period in type II diabetic patients with a clinical diagnosis of diabetic kidney disease. BAY1142524 or placebo will be given on top of evidence-based standard of care for diabetic kidney disease. Primary objective is the analysis of first signs of efficacy as determined by favourable changes in urinary albumin creatinine ratio. Secondary objective is the analysis of safety and tolerability as evidenced by the incidence and severity of adverse events. 64 valid patients have to complete treatment with verum and 32 valid patients have to complete treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus and a clinical diagnosis of diabetic kidney disease (DKD) (as judged by the investigator) who have finished their up-titration with an angiotensin receptor blocker (ARB) or an ACEI (angiotensin-converting enzyme inhibitor) to their maximum tolerated dose at least 3 months prior to the screening visit, whereby the maximum tolerated dose has to be at least as high as the minimal recommended dose of an ARB or ACEI according to local and/or international guidelines. Patients have to be treated with an ARB or ACEI, but not with both simultaneously, without any adjustments to this therapy for at least 4 weeks prior to the screening visit.
* UACR >50 mg/g and <3000 mg/g in 2 out of 3 consecutive morning void samples at the screening and the baseline visit
* estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m*2 and <90 mL/min/1.73 m*2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) at the screening visit and the baseline visit

Exclusion Criteria:

* Non-DKD if it is the main diagnosis contributory to chronic kidney disease (CKD), as judged by the investigator
* Known bilateral clinical relevant renal artery stenosis (>75%)
* New York Heart Association (NYHA) Class IV
* Acute kidney injury or dialysis within the last 3 months before the screening visit
* Renal replacement therapy during study conduct
* Renal allograft in place or a scheduled kidney transplant during study conduct
* Stroke, transient ischemic cerebral attack, acute coronary syndrome, or hospitalization for heart failure in the last 3 months prior to screening visit
* Clinically relevant hepatic dysfunction
* Uncontrolled hypertension as evidenced by systolic blood pressure >160 mmHg, diastolic blood pressure >100 mmHg (mean of triplicate values at the screening or baseline visit)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Change in urinary albumin to creatinine ratio (UACR) | Baseline and at 6 months
  The ratio of albumin to creatinin will be determined in first morning void urine at baseline (before treatment start) and after 6 months of treatment

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse event | From first intake of study drug up to 3 days after last administration of study drug
Number of patients with serious adverse events | From first intake of study drug up to 3 days after last administration of study drug

CONTACTS AND LOCATIONS:
Locations (27):
- Bulgaria (3):
  - Med Centre Diamedical 2013, Dimitrovgrad
  - MCOMH Preventsia-2000, Stara Zagora
  - Med. Center Equita, Varna
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Nordsjællands Hospital, Hillerød
- Finland (4):
  - Pihlajalinna ITE Kuopio, Kuopio
  - Terveystalo Oulu, Oulu
  - TAYS TKI Keskus Tutkimusvastaanotto, Tampere
  - Turun yliopistollinen keskussairaala, kantasairaala, Turku
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Edith Wolfson Medical Center, Holon
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - The Nazareth Trust Hospital EMMS, Nazareth
  - DMC - Diabetes Medical Center, Tel Aviv
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (4):
  - IRCCS Casa Sollievo della Sofferenza, Foggia, Apulia
  - A.O.U. Policlinico Federico II Napoli, Napoli, Campania
  - Univ. Alma Mater - Dip. Medicina Spec, Diagnostica e Sperim, Bologna, Emilia-Romagna
  - A.O.U. di Padova, Padua, Veneto
- Spain (3):
  - Complexo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital Fundació Puigvert, Barcelona
- Sweden (4):
  - Centralsjukhuset Kristianstad, Kristianstad
  - Universitetssjukhuset Örebro, Örebro
  - Akardo MedSite AB, Stockholm
  - S3 Clinical Research Centers, Vällingby

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/